CLINICAL TRIAL: NCT01571128
Title: Gender-Specific Combination HIV Prevention for Youth in High Burden Settings (MP3-Youth)
Acronym: MP3-Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: University of Nairobi (Other); Impact Research & Development Organization (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01AI094607-1; 1R01AI094607 (NIH)
Record Dates: First submitted 2012-02-08; First posted 2012-04-05 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2018-09

CONDITIONS: HIV; Adolescent Behavior; Gender
Keywords: HIV; Prevention & Control; Intervention Studies; Adolescent; Gender; Combination prevention; Pre-Exposure Prophylaxis; Cash Transfer; Medical Male Circumcision; HIV Testing; Mobile Health
MeSH Terms: conditions — Adolescent Behavior; Coitus | interventions — Condoms; Contraception; Family Planning Services; Pre-Exposure Prophylaxis; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Tenofovir; Economics, Behavioral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Male-Specific Intervention Package (Experimental): Gender-specific interventions targeted specifically for boys offered in an integrated services delivery modality. Cross-Sectional Arm.
  Interventions: Other: Male-Specific Intervention Package
- Female-Specific Intervention Package (Experimental): Gender-specific interventions targeted specifically for girls offered in an integrated services delivery modality. Cross-Sectional Arm.
  Interventions: Other: Female-Specific Intervention Package
- HIV Positive Cohort (Males and Females) (No Intervention): Behavioral data on HIV positive youth. Longitudinal Arm.
- Pre-Exposure Prophylaxis (Females) (Experimental): PrEP adherence and feasibility. Longitudinal Arm.
  Interventions: Drug: Pre-Exposure Prophylaxis (Females)
- Cash Transfer Cohort (Females) (Experimental): School attendance, behavioral data, and feasibility. Longitudinal Arm
  Interventions: Behavioral: Cash Transfer Cohort (Females)

INTERVENTIONS:
Other: Male-Specific Intervention Package — Combination HIV Prevention: Male-Specific Intervention Package at the Mobile Health events and longitudinal follow up of cohorts.
  Other Names: HIV Counseling and Testing (HTC); Facilitated linkage to care for HIV+: ART/PMTCT; Condoms; Voluntary Medical Male Circumcision (VMMC)
  Arms: Male-Specific Intervention Package
Other: Female-Specific Intervention Package — Combination HIV Prevention: Female-Specific Intervention Package at the Mobile Health events and longitudinal follow up of cohorts.
  Other Names: HIV Counseling and Testing (HTC); Facilitated linkage to care for HIV+: ART/PMTCT; Contraception/Family Planning (FP); Pre-exposure Prophylaxis (PrEP); Conditional Cash Transfer (CCT)
  Arms: Female-Specific Intervention Package
Drug: Pre-Exposure Prophylaxis (Females) — Females 18-24 who are out of school.
  Other Names: Truvada; Emtricitabine; Tenofovir disoproxil fumarate
  Arms: Pre-Exposure Prophylaxis (Females)
Behavioral: Cash Transfer Cohort (Females) — Cash transfer for females (and their parents) who are aged 15-24 and enrolled in school.
  Other Names: Behavioral Economics; Conditional Cash Transfer
  Arms: Cash Transfer Cohort (Females)

SUMMARY:
MP3 Youth is a pilot study to evaluate the feasibility and acceptability of a gender-specific combination HIV prevention package for youth (aged 15-24) in high burden settings. The study aims to pilot a combination package of gender-specific interventions in western Kenya in a mobile health delivery format using integrated services delivery.

DETAILED DESCRIPTION:
The MP3-Youth study will provide critical information for design and evaluation of combination HIV prevention intervention packages that are sensitive to gender-specific risks among this most-at-risk population in high-HIV burden African settings. Our team of biobehavioral and clinical scientists, mathematical modelers, and trial design specialists will:

Aim 1: Identify gender (sex)-specific drivers of HIV acquisition risk, including pregnancy among females, for youth in sub-Saharan Africa, and interventions to best address those risks.

Aim 2: Conduct mathematical modeling to select optimal combination intervention package components and to assess potential population-level impact.

Aim 3: In partnership with a highly-productive nongovernmental organization (NGO) that is delivering PEPFAR-funded HIV prevention services, develop and pilot a combination HIV prevention package specific for female and for male youth - 'MP3-Youth' - in Nyanza Province, Kenya.

Aim 4: Design a phase IV study protocol for testing the effectiveness of a gender-specific youth HIV prevention package in sub-Saharan Africa. We will disseminate these research protocol recommendations, and study instruments including the mathematical modeling tool, as a combination prevention intervention research toolkit.

Design: Study activities comprise systematic review and meta-analysis of the HIV prevention literature for youth in sub-Saharan Africa; development of a mathematical modeling tool; and a community-based HIV combination prevention pilot that will take place in western Kenya. These activities will culminate in a testable combination HIV prevention trial protocol for youth, which is the main study deliverable.

Population: Aim 1: Focus groups will be held with male and female youth, parents, teachers, religious and community leaders. Aim 3: Pilot study will include male and female youths (ages 15-24) from Nyanza Province, Kenya.

Deliverables: Study deliverables include selection procedures for a population-specific combination HIV prevention package; measurement instruments, mobile prevention delivery protocols, mathematical modeling tools, and a testable study trial protocol. The entire MP3-Youth Package will be placed on a web site for open access.

ELIGIBILITY:
Inclusion Criteria:

* Any male or female between the ages of 15-24.
* Able to understand spoken English or Kiswahili or Dholuo.
* Willing to give informed consent or if younger than 18 years of age has a parent or guardian willing to provide consent in addition to the minor's assent
* Willing to be tested for HIV.
* Willing to get participant ID based on biometric finger scan.

Exclusion Criteria:

* Any male or female younger than 15 or older than 24.
* Unable to understand spoken English, or Kiswahili or Dholuo.
* If under 18 and not an emancipated minor, unable to get parental consent.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1215 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-03-23 (Actual); Study Completion 2016-03-23 (Actual)

PRIMARY OUTCOMES:
Intervention Uptake (acceptability) and Coverage (feasibility) | 6 months
  * Coverage: The proportion of youth in the community who attend each mobile event (estimated from youth population denominator)
  * Enrollment: The number of participants who consent to being enrolled in the study during each mobile event.
  * Uptake: The number of participants who choose one or more components of their tailored combination package (and which components).
  * Intervention Acceptability: Satisfaction with mobile event services

SECONDARY OUTCOMES:
Adherence to medication (HIV+ and PrEP cohort participants only) over 12 months | 12 months
  * Adherence to once daily Truvada (PrEP) among HIV-uninfected eligible females and patterns of adherence and sexual HIV acquisition risk exposure (PrEP cohort participants only). Measured by self-report, eCAPs, and clinical assessments; monthly for first 6 months and every 3 months for the following 6 months and DBS for analysis of TFV/FTC: TFV-DP/FTC-TP at months 2 and 9.
  * Adherence to ART for positives (HIV+ cohort participants only). Measured by self-report monthly SMS: 0, 3, 6,9,12 months). POC CD4 and baseline viral load by dried blood spot will be measured at mobile event baseline and repeated at 12 months.

OTHER OUTCOMES:
Feasibility of administering cash transfer to keep girls in school | 12 months
  Conditional Cash Transfer to reduce HIV risk by staying in school.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Inwani, MD, MPH, Principal Investigator — Kenyatta National Hospital: University of Nairobi, Kenya; Ann Kurth, PhD, CNM, Principal Investigator — New York University; Jasmine Buttolph, MPH, Study Director — New York University
Locations (3):
- New York University, New York, New York, United States
- Kenya (2):
  - Impact Research and Development Organization, Kisumu
  - University of Nairobi, Nairobi

REFERENCES:
- [Derived] Buttolph J, Inwani I, Agot K, Cleland CM, Cherutich P, Kiarie JN, Osoti A, Celum CL, Baeten JM, Nduati R, Kinuthia J, Hallett TB, Alsallaq R, Kurth AE. Gender-Specific Combination HIV Prevention for Youth in High-Burden Settings: The MP3 Youth Observational Pilot Study Protocol. JMIR Res Protoc. 2017 Mar 8;6(3):e22. doi: 10.2196/resprot.5833. PMID 28274904